CLINICAL TRIAL: NCT03618771
Title: The Functional Outcomes and Stability of Total Knee Replacement Design Concepts
Brief Title: A Functional Comparison of Two TKR Designs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Manchester University NHS Foundation Trust (Other Government)
Collaborators: Medacta International SA (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: B00116
Record Dates: First submitted 2018-06-19; First posted 2018-08-07 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Knee Osteoarthritis
Keywords: Total Knee Arthroplasty; Osteoarthritis; Stability; Knee; Functional Outcome; Gait; Biomechanics
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis | interventions — Arthroplasty, Replacement, Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Medacta GMK Sphere (Experimental): Half of the patients will be implanted with the Medacta GMK Sphere total knee arthroplasty
  Interventions: Device: Total knee arthroplasty
- DePuy Synthes Attune (Experimental): Half of the patients will be implanted with the DePuy Attune total knee arthroplasty
  Interventions: Device: Total knee arthroplasty

INTERVENTIONS:
Device: Total knee arthroplasty — Parts of the knee joint diseased by osteoarthritis are replaced by metal and plastic prostheses.
  Other Names: Medacta GMK Sphere Implant; DePuy Synthes Attune Implant

SUMMARY:
Total knee replacement (TKR) is an established treatment for knee osteoarthritis and leads to a satisfactory outcome in over 75% of patients. However, up to 25% of patients are not entirely satisfied with their TKR. Patient dissatisfaction has been associated with inadequate functional outcome, especially during negotiation of stairs and slopes. This phenomenon, known as mid-flexion instability, is believed to be caused by excessive anterior-posterior motion of the implant during activities of daily living. This is characterised as a perception that the replaced knee is unsteady during certain tasks.

This study will compare the functional outcome of two implants that have been designed to provide patients with a functionally stable knee throughout its range of motion. The different design roles in preventing implant-related mid-flexion instability remain unknown. The functional outcome and stability of these implants will be tested non-invasively with 3D motion capture technology.

DETAILED DESCRIPTION:
This study will compare the functional outcome of two implants that have been designed to provide patients with a functionally stable knee throughout its range of motion. The different design roles in preventing implant-related mid-flexion instability remain unknown.

The Medacta GMK-Sphere implant consists of a fully congruent medial compartment which allows freedom of movement in the lateral compartment. Both femoral and tibial components are also available in a range of 13 sizes, allowing the surgeon to find a 'best fit' for each patient. These design features are aimed to mimic the movement of a natural healthy knee, potentially preventing implant-related mid-flexion instability.

The DePuy Synthes Attune implant design aims to provide patients with optimal functional outcome. The femoral component of this implant has a gradually reducing radius, and the tibial component an S-shaped post-cam mechanism. These features are designed to facilitate smooth movement and stability during flexion.

The comparative functional outcomes and stability in gait, and other activities of daily living has not been established for the two different TKR design concepts. Functional assessments will be carried out on TKR patients pre- and post-operatively. These assessments will non-invasively quantify the knee's stability, range of motion, strength as well as walking kinematics using 3D motion capture technology. As mid-flexion instability is most notable during downhill walking, patients will be required to walk downhill on a treadmill as part of this study, to better investigate the phenomenon of mid-flexion knee instability.

This study will not involve any invasive procedure in addition to the standard of care. As such, the research burden is minimal. The main ethical issue may be that patients will not be randomised into one of the two proposed groups.

Patients will receive either the GMK-Sphere implant or the Attune implant according to their surgeon's usual practice. Surgeons who specialise in the GMK-Sphere implant will only implant the GMK-Sphere for this study, and surgeons who specialise in the Attune implant will only implant the Attune. This allows surgeons to undertake the prosthesis with which they are expert, and also limit potential surgical error in the case of surgeons having to randomise patients to different designs on the same list.

Patients will be seen by the trial team on 3 separate occasions:

1. Routine pre-admission clinic: Recruitment, collection of patient information and questionnaire data and completion of pre-operative physical tests (including gait analysis with 3D motion capture technology)
2. Routine post-operation clinic: Six-weeks post-operative physical tests (including gait analysis with 3D motion capture technology) and questionnaire data
3. Annual post-operation clinic: 1-year post-operative physical tests (including gait analysis with 3D motion capture technology) and questionnaire data

   Collection of baseline data during pre-admission clinic (standard care except physical tests):
   * Descriptive: Patient demographics (sex, age, height, mass, BMI), diagnosis, pattern of OA, medical co-morbidity
   * Questionnaire Data

     * Oxford Knee Score - A joint specific questionnaire which asks patients on the level of pain and function they believe to have in their affected knee.
     * EQ5D - A questionnaire on patients' perception of their overall health. It contains a visual analogue scale where patients have to choose on a scale of 0-100 how well they believe their general health to be.
     * SF12 - A general Quality of Life score. It has mental and physical components.
     * Forgotten Joint Score - This asks questions not covered in the OKS on patient perception of their knee that are important to know following TKA. It focuses on other aspects of outcome other than joint pain and function.
     * Expectation questionnaire - This asks what the patients expect from the surgery. The investigators use this to gauge whether patients are expecting to achieve too much or too little post-op. This is important for understanding post-operative patient satisfaction.

   All questionnaires ask different questions (although there is some overlap). Together, they give an overall view of the patients' perception of their general health and knee specific problems. As such, they are all deemed necessary for this investigation.

   There are separate scoring sheets for these subjective quantitative scores. The results are typically presented as a Mean ± SD score for each questionnaire (provided the data is normally distributed). All are valid in the English language.

   • Non-invasive Physical Tests: Range of knee movement, knee muscular strength, lower limb kinematics during level (0°)- and downhill (7.5°)-walking

   Collection of follow-up measures by trial team between operation and post-operative visit (standard care):

   • Surgical complications

   Collection of data during routine follow-up clinics:

6 weeks post-operation (standard care except physical tests):

* Questionnaire Data: Oxford Knee Score, SF12, EQ5D, Forgotten Joint Score
* Non-invasive Physical Tests: Range of knee movement, knee muscular strength, lower limb kinematics during level (0°)- and downhill (7.5°)-walking

  12 weeks post-operation (standard care):
* Descriptive: Radiographic measurement of alignment (Non-invasive)

  1 year post-operation (standard care except physical tests):
* Questionnaire Data: Oxford Knee Score, SF12, EQ5D, Forgotten Joint Score, Satisfaction questionnaire
* Descriptive: Late complications
* Non-invasive Physical Tests: Range of knee movement, knee muscular strength, lower limb kinematics during level (0°)- and downhill (7.5°)-walking

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of osteoarthritis of the knee which is sufficiently symptomatic to require knee arthroplasty as assessed by their consultant orthopaedic surgeon

Exclusion Criteria:

* Inflammatory arthropathy
* Patients requiring bone augmentation
* Patients with collateral ligament incompetence
* Valgus deformity >5 degrees.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 2019-02-06 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Gait Kinematics at 1-Year | Change from baseline at 1-Year
  Gait of patients will be analysed pre-operatively, six-weeks post-operatively, and 1-year post-operatively by 3D motion capture technology. The change measured over time at 1-year will be the primary outcome.

SECONDARY OUTCOMES:
Patient Satisfaction (Pain/Hospital experience/functional ability/Surgery expectations) | 1 year post-operatively
  Patient satisfaction will be reported using a scale on a questionnaire which asks six questions on how happy patients were with their hospital experience/level of pain/functional ability post-operatively. The questionnaire also asks whether their expectations were met. The two satisfaction questions are answered on a scale of 'Very Satisfied/Satisfied/Unsure/Dissatisfied' by ticking the appropriate box. The four questions based on patient expectation are scored on a scale of 'Excellent/Good/Unsure/Poor' by ticking the appropriate box.
Oxford Knee Score (Patient reported outcome measure of pain and function) | Pre-operatively
  A joint specific questionnaire which asks patients on the level of pain and function they believe to have in their affected knee (taking into consideration the past 4 weeks only). The questionnaire consists of 12 questions. Five of the questions are pain related, and seven are aimed at function. Each question has 5 options and is scored from 0-4, with 4 being the best and 0 being the worst pain/function. The best score is therefore 48 (no pain/good function), and the worst score is 0 (pain and poor function).
Oxford Knee Score (Patient reported outcome measure of pain and function) | 6 weeks post-operatively
  A joint specific questionnaire which asks patients on the level of pain and function they believe to have in their affected knee (taking into consideration the past 4 weeks only). The questionnaire consists of 12 questions. Five of the questions are pain related, and seven are aimed at function. Each question has 5 options and is scored from 0-4, with 4 being the best and 0 being the worst pain/function. The best score is therefore 48 (no pain/good function), and the worst score is 0 (pain and poor function).
Oxford Knee Score (Patient reported outcome measure of pain and function) | 1 year post-operatively
  A joint specific questionnaire which asks patients on the level of pain and function they believe to have in their affected knee (taking into consideration the past 4 weeks only). The questionnaire consists of 12 questions. Five of the questions are pain related, and seven are aimed at function. Each question has 5 options and is scored from 0-4, with 4 being the best and 0 being the worst pain/function. The best score is therefore 48 (no pain/good function), and the worst score is 0 (pain and poor function).
EuroQol-5 Dimensions (EQ-5D) (Patient reported outcome measure of patients' perception of their overall health) | Pre-operatively
  A questionnaire on patients' perception of their overall health. The questionnaire focuses on generic health in 5 dimensions: Mobility, self-care, pain or discomfort, anxiety or depression and usual activities (including work, housework, leisure, family, and study). The questions are scored using an algorithm; the result of which relates to the health status of the patient. This score ranges between 0 (equivalent to death) to 1 (equivalent to full health). It also contains a visual analogue scale where patients have to choose on a scale of 0-100 how well they believe their general health to be on that particular day, where 0 is the worst health imaginable and 100 is the best health imaginable.
EuroQol-5 Dimensions (EQ-5D) (Patient reported outcome measure of patients' perception of their overall health) | 6 weeks post-operatively
  A questionnaire on patients' perception of their overall health. The questionnaire focuses on generic health in 5 dimensions: Mobility, self-care, pain or discomfort, anxiety or depression and usual activities (including work, housework, leisure, family, and study). The questions are scored using an algorithm; the result of which relates to the health status of the patient. This score ranges between 0 (equivalent to death) to 1 (equivalent to full health). It also contains a visual analogue scale where patients have to choose on a scale of 0-100 how well they believe their general health to be on that particular day, where 0 is the worst health imaginable and 100 is the best health imaginable.
EuroQol-5 Dimensions (EQ-5D) (Patient reported outcome measure of patients' perception of their overall health) | 1 year post-operatively
  A questionnaire on patients' perception of their overall health. The questionnaire focuses on generic health in 5 dimensions: Mobility, self-care, pain or discomfort, anxiety or depression and usual activities (including work, housework, leisure, family, and study). The questions are scored using an algorithm; the result of which relates to the health status of the patient. This score ranges between 0 (equivalent to death) to 1 (equivalent to full health). It also contains a visual analogue scale where patients have to choose on a scale of 0-100 how well they believe their general health to be on that particular day, where 0 is the worst health imaginable and 100 is the best health imaginable.
Short Form-12 (SF-12) (Patient reported outcome measure of general quality of life) | Pre-operatively
  A general Quality of Life score with 12 questions. It has mental and physical components which are scored from the same questions, using different algorithms. Each question is multiple choice, and the patient must tick one answer. Each answer corresponds to a standardised value, which is used in two algorithms to generate an overall score. One score is for the mental component and one is for the physical component. The physical standardized values are summed across all 12 items. 56.57706 is added to the sum to create the SF-12 physical score. 60.75781 is added to sum create the SF-12 mental score. Higher overall scores are better than lower scores.
Short Form-12 (SF-12) (Patient reported outcome measure of general quality of life) | 6 weeks post-operatively
  A general Quality of Life score with 12 questions. It has mental and physical components which are scored from the same questions, using different algorithms. Each question is multiple choice, and the patient must tick one answer. Each answer corresponds to a standardised value, which is used in two algorithms to generate an overall score. One score is for the mental component and one is for the physical component. The physical standardized values are summed across all 12 items. 56.57706 is added to the sum to create the SF-12 physical score. 60.75781 is added to sum create the SF-12 mental score. Higher overall scores are better than lower scores.
Short Form-12 (SF-12) (Patient reported outcome measure of general quality of life) | 1 year post-operatively
  A general Quality of Life score with 12 questions. It has mental and physical components which are scored from the same questions, using different algorithms. Each question is multiple choice, and the patient must tick one answer. Each answer corresponds to a standardised value, which is used in two algorithms to generate an overall score. One score is for the mental component and one is for the physical component. The physical standardized values are summed across all 12 items. 56.57706 is added to the sum to create the SF-12 physical score. 60.75781 is added to sum create the SF-12 mental score. Higher overall scores are better than lower scores.
Forgotten Joint Score (Patient reported outcome measure of awareness of knee) | Pre-operatively
  This asks questions not covered in the OKS on patient perception of their knee that are important to know following TKA. It focuses on other aspects of outcome other than joint pain and function. There are 12 questions in total, each starting with 'Are you aware of your knee joint...' followed by a daily situation such as driving/lying in bed etc. Each question has a possible of 5 answers: Never/Almost Never/Seldom/Sometimes/Mostly. Every question is scored 1 (never) to 5 (mostly) according to the selected response categories. Thus, the raw score ranges from 12 to 60. The raw score is linearly transformed to a 0-100 scale and then reversed to obtain the final score. For the final Forgotten Joint Score -12 a high score indicates good outcome.
Forgotten Joint Score (Patient reported outcome measure of awareness of knee) | 6 weeks post-operatively
  This asks questions not covered in the OKS on patient perception of their knee that are important to know following TKA. It focuses on other aspects of outcome other than joint pain and function. There are 12 questions in total, each starting with 'Are you aware of your knee joint...' followed by a daily situation such as driving/lying in bed etc. Each question has a possible of 5 answers: Never/Almost Never/Seldom/Sometimes/Mostly. Every question is scored 1 (never) to 5 (mostly) according to the selected response categories. Thus, the raw score ranges from 12 to 60. The raw score is linearly transformed to a 0-100 scale and then reversed to obtain the final score. For the final Forgotten Joint Score -12 a high score indicates good outcome.
Forgotten Joint Score (Patient reported outcome measure of awareness of knee) | 1 year post-operatively
  This asks questions not covered in the OKS on patient perception of their knee that are important to know following TKA. It focuses on other aspects of outcome other than joint pain and function. There are 12 questions in total, each starting with 'Are you aware of your knee joint...' followed by a daily situation such as driving/lying in bed etc. Each question has a possible of 5 answers: Never/Almost Never/Seldom/Sometimes/Mostly. Every question is scored 1 (never) to 5 (mostly) according to the selected response categories. Thus, the raw score ranges from 12 to 60. The raw score is linearly transformed to a 0-100 scale and then reversed to obtain the final score. For the final Forgotten Joint Score -12 a high score indicates good outcome.
Knee Strength | Pre-operatively
  Knee strength in Newton meters will be assessed using motion capture technology and a dynamometer
Knee Strength | 6 weeks post-operatively
  Knee strength in Newton meters will be assessed using a dynamometer.
Knee Strength | 1 year post-operatively
  Knee strength in Newton meters will be assessed using a dynamometer.
Knee range of motion | Pre-operatively
  Knee range of motion in degrees will be assessed using motion capture technology
Knee range of motion | 6 weeks post-operatively
  Knee range of motion in degrees will be assessed using motion capture technology
Knee range of motion | 1 year post-operatively
  Knee range of motion in degrees will be assessed using motion capture technology.

CONTACTS AND LOCATIONS:
Overall Officials: Leela C Biant, FRCSEd Tr & Orth, Principal Investigator — University of Manchester
Locations (1):
- Trafford General Hospital, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No